CLINICAL TRIAL: NCT05720624
Title: Pharmacodynamic Analyses of Metabolic Agents Following Brain Radiation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding issues
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MC220708; NCI-2022-10632 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-003783 (Other: Mayo Clinic in Rochester); MC220708 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-01-17; First posted 2023-02-09 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Malignant Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Oxaloacetic Acid; Practice Guidelines as Topic; Standard of Care; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort I, Arm A (standard of care therapy) (Active Comparator): Patients in Cohort I, Arm A receive standard of care therapy. Patients also undergo MRS imaging, collection of CSF, and collection of blood on study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Questionnaire Administration
- Cohort I, Arm B ( standard of care therapy, AEO) (Experimental): Patients in Cohort I, Arm B receive standard of care therapy and receive AEO PO BID for 1 month on study. Patients also undergo MRS imaging, collection of CSF, and collection of blood on study.
  Interventions: Drug: Anhydrous Enol-oxaloacetate; Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Questionnaire Administration
- Cohort II, Arm A (standard of care therapy) (Active Comparator): Patients in Cohort II, Arm A receive standard of care therapy. Patients also undergo MRS imaging, collection of CSF, and collection of blood on study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Questionnaire Administration
- Cohort II, Arm B (standard of care therapy, AEO) (Experimental): Patients in Cohort II, Arm B receive standard of care therapy and receive AEO PO BID for 3 months on study. Patients also undergo MRS imaging, collection of CSF, and collection of blood on study.
  Interventions: Drug: Anhydrous Enol-oxaloacetate; Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Spectroscopic Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Anhydrous Enol-oxaloacetate — Given PO
  Other Names: AEO; OXALOACETIC ACID
  Arms: Cohort I, Arm B ( standard of care therapy, AEO); Cohort II, Arm B (standard of care therapy, AEO)
Other: Best Practice — Receive standard of care therapy
  Other Names: standard of care; standard therapy
Procedure: Biospecimen Collection — Undergo collection of CSF and blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRS imaging
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; MS; Proton Magnetic Resonance Spectroscopic Imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the impact of taking drugs (agents) that target altered brain metabolism following standard of care brain radiotherapy. Radiotherapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. However, radiotherapy can also cause harmful effects to normal brain functioning. One drug, called anhydrous enol-oxaloacetate (AEO), has previously been studied in ischemic stroke, Alzheimer's disease, Parkinson's disease, and glioma. Drugs such as AEO may help preserve or restore healthy brain function after brain radiotherapy compared to the standard practice which consists of no drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of serial cerebrospinal fluid (CSF) assessments to evaluate the pharmacodynamic impact of agents targeting radiation-induced biology administered following completion of brain radiation.

SECONDARY OBJECTIVE:

I. Assess the safety of study drug(s) as quantified by dose-limiting toxicities.

CORRELATIVE RESEARCH OBJECTIVES:

I. Investigate the relationship of the global CSF metabolome with magnetic resonance spectroscopy metabolite profile.

II. Investigate the relationship between brain radiation dose/volume and metabolic alterations in CSF.

III. Investigate the impact of metabolic therapy on early cognitive effects of radiotherapy in patients with brain tumors.

IV. Utilize paired blood samples to investigate association between the CSF and systemic metabolome.

V. Utilize paired stool samples to investigate association between the blood and CSF metabolome with the gastrointestinal microbiome.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I (EARLY POST-RADIATION): Patients within Cohort I are assigned to 1 of 2 arms.

ARM A: Patients receive standard of care therapy.

ARM B: Patients receive standard of care therapy and receive AEO orally (PO) two times daily (BID) for 1 month on study.

COHORT II (DELAYED POST-RADIATION): Patients within Cohort II are assigned to 1 of 2 arms.

ARM A: Patients receive standard of care therapy.

ARM B: Patients receive standard of care therapy and receive AEO PO BID for 3 months on study.

Patients in all cohorts and arms also undergo magnetic resonance spectroscopy (MRS) imaging, collection of cerebrospinal fluid (CSF), and collection of blood on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Radiographic evidence or histopathologic confirmation of central nervous system (CNS) malignancy, with or without prior resection.
* Planned (cohort 1) or completed (cohort 2) fractionated brain radiation. The therapeutic brain radiation treatment volume should exceed 30 cubic cm, including the volume of brain tissue occupied by infiltrative disease. Volume occupied by solid non-infiltrative disease (e.g. meningioma, metastatic disease, cystic cavity, resection cavity), should be excluded from the estimated treatment volume.
* Provide written informed consent for the current study and the Neuro-oncology biorepository for archiving of CSF and blood samples collected on this protocol.
* Expected survival >6 months and Karnofsky performance status >= 60.
* Willing and able to adhere with the protocol for the duration of the study including undergoing treatment and scheduled visits, and examinations.
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) <3 x upper limit of normal (ULN) (=< 5 x ULN for patients with baseline liver disease).
* Serum creatinine =< 1.5 mg/dL.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Willingness to provide mandatory CSF and blood and able to undergo magnetic resonance spectroscopy (MRS)/magnetic resonance imaging (MRI) with gadolinium.
* Male and female patients of childbearing potential must agree to use a dual method of contraception (a highly effective method of contraception in conjunction with barrier contraception) consistently and correctly from the first dose of study drug (Arm B only) until 90 days after the last dose of study drug.

Exclusion Criteria:

* Uncontrolled and/or intercurrent illness which limits safety of or compliance to study proceedings.
* Vulnerable populations: pregnant or nursing women (Arm B exempt), prisoners, mentally handicapped.
* Patients with recurrent brain tumor after prior radiation.
* Cohort 1 only: History of prior brain radiation, with prior cumulative target radiation treatment volume exceeding 2 cubic centimeters.
* Patients who do not have an implanted CSF access device (who would thus require multiple lumbar punctures [LPs] for participation) should be excluded if they have any contra-indication to lumbar puncture. This includes but is not limited to obstructive hydrocephalus or posterior fossa mass or cerebral edema that could increase the risk of brain herniation.
* Patients who do not have an implanted CSF device and are on anti-platelet therapy (other than Aspirin which is considered low risk) or anticoagulation (coumadin, Eliquis) must discontinue these prior to each lumbar puncture to participate. Patients unwilling or unable to safely do so should not be enrolled.
* Participants who are unable to swallow tablets or who are at risk for impaired absorption of oral medication. NOTE: This includes but not limited to, refractory vomiting, gastric resection/bypass, and duodenal/jejunal resection.
* Patients with recent (<3 months [mo]) administration of, or known hypersensitivity or allergy to any active study drug currently available for randomization (initially oxaloacetate).
* Current use of resveratrol, CoQ10 (coenzyme Q10), coconut oil/other medium chain triglyceride-containing (i.e. Axona) supplements, or curcumin will be excluded unless willing to discontinue them 14 days prior to the start of baseline visits and remain off for study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of completing serial cerebrospinal fluid (CSF) collections for pharmacodynamic analyses. | Up to 3 months
  Successful collection of at least 1cc of CSF at each of 3 timepoints with successful quantification of glutamate and lactate from each sample.

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (AEs) related to oxaloacetate following brain radiation (Arms B and Future Arms) | Up to 3 months
  To assess the safety and tolerability of the study drug(s). Safety will be assessed in that the study drug will not have a Common Terminology Criteria for Adverse Events (CTCAE) (version [v] 5.0) grade >3 in >20% of participants. Tolerability will be assessed in that >60% of participants are able to complete the initial 28-day study treatment period without AE precluding continuation of study drug (even if not CTCAE >3).

CONTACTS AND LOCATIONS:
Overall Officials: Terence C. Burns, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials